CLINICAL TRIAL: NCT00155571
Title: The Occurrence of Periopathogens in Betel-Nut Chewers and the Effects of Areca-Nut on Periopathogens
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 14881; NSC-90-2314-B-002-357
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2001-01

CONDITIONS: Periodontitis
Keywords: betel nut; periodontitis; periodontal microbiology
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Periodontal disease is considered to be an infection disease. Recent evidence supported the role of smoking as a potent risk factor for the development of periodontal disease. However, the effect of another oral habit, betel quid chewing on periodontal tissues has not been well determined. The purpose of the present study is to analysis the role of bacteria on the periodontium in the betel quid chewers. Plaque samples will be collected from betel quid chewers and the occurrence of periodotopathogens will be analyzed Since most chewers also smokers, plaque samples from age matched smokers but not betel chewers and non-smokers will analysis for comparison. An in vitro test is also performed to evaluate whether the extract has a direct inhibitory effect on common periodontal pathogens, such as Porphyromoans gingivalis, Bacteroides forsythus, Actinobacillus actinomycetemcomitans.

DETAILED DESCRIPTION:
Periodontal disease is considered to be an infection disease. Specific microorganisms especially the gram-negative anaerobic bacteria gain predominance in periodontal pockets and challenge the host. Lipopolysaccharides of the bacteria and other virulence factors will interact with macrophages and active cells to synthesis large quantities of IL-1, TNF, PgE2 and matrix metalloproteinases and lead to the degradation of the collagen and bone destruction. It has been shown that the genetic or environmental factors can modulate the initiation and progression of periodontal disease. Recent evidence supported the role of smoking as a potent risk factor for the development of periodontal disease. However, the effect of another oral habit, betel quid chewing on periodontal tissues has not been well determined. Earlier epidemiological studies have shown a detrimental effect on periodontal tissues. Higher prevalence of periodontal disease among betel chewers than among non-chewers was found, even when subgroups of similar oral hygiene were compared. In vitro studies also support the nut extract has a cytopathologic effects on gingival fibroblast. The extract or the major betel nut alkaloid, arecoline, can inhibit the growth, attachment and matrix protein synthesis of gingival fibroblast. Study also showed that ripe and tender extract can reduce the antibacterial activity of neutrophils in vitro. However, most earlier epidemiological studies did not adjust the potentially confounding variables such as age, socioeconomic status, oral hygiene. Besides, most chewers are also smokers and drinkers, whether the higher periodontal index may contribute from the smoking habit, or betel quid chewing or the combination of both habits cannot be determined. Conversely, it is also found that the betel nut has an antibacterial properties and prolonged exposure can suppress the salivary organisms. It is also used for treating bleeding gums in ancient Indian medicine. Inhibitory effect on Streptococcus mutans, Streptococcus salivarius, Fusbobacerium nucleatum was shown, but there are no any data concerning the effect on the periodontal pathogens. Since the challenge of the bacteria is essential to initiate the disease process, the presence of more virulence types of plaque bacteria may increase the risk and the rate of progression of periodontal disease. It is not known whether the extract can affect the composition of the dental plaque through changing the oral ecology such as the pH value of the saliva, a direct inhibitory effect on the periodontal microorganism or through inhibiting the colonization of the Streptococcus, and then prevent the further succession of another bacterial complex. The purpose of the present study is to analysis the role of bacteria on the periodontium in the betel quid chewers. Plaque samples will be collected from betel quid chewers and the occurrence of periodotopathogens will be analyzed Since most chewers also smokers, plaque samples from age matched smokers but not betel chewers and non-smokers will analysis for comparison. An in vitro test is also performed to evaluate whether the extract has a direct inhibitory effect on common periodontal pathogens, such as Porphyromoans gingivalis, Bacteroides forsythus, Actinobacillus actinomycetemcomitans.

ELIGIBILITY:
Inclusion Criteria:

- Smoker/periodontitis Betel nut chewer/periodontitis Healthy

Exclusion Criteria:

systemic disease

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Man-ying Wang, DDS, MS, Principal Investigator — Department of Periodontics, National Taiwan University Hospital
Locations (1):
- National Taiwan Univerity hospital, Dawan, Taiwan